CLINICAL TRIAL: NCT00823628
Title: Comparison of Contrast-medium Induced Nephrotoxicity Between Iodixanol and Iopromide in Patients With Renal Insufficiency Undergoing Coronary Angiography
Brief Title: Contrast-medium Induced Nephrotoxicity in Patients Undergoing Coronary Angiography - Iodixanol Versus Iopromide
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Tae-Jin Youn / Associate professor, Cardiovascular Center, Seoul National University Bundang Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: B-0902/069-003
Record Dates: First submitted 2009-01-14; First posted 2009-01-15 (Estimated); Last update posted 2010-07-07 (Estimated); Status verified 2009-04

CONDITIONS: Chronic Renal Insufficiency; Coronary Angiography
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Contrast Media; iopromide; iodixanol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- iopromide (Active Comparator)
  Interventions: Drug: contrast agent (iopromide)
- iodixanol (Experimental)
  Interventions: Drug: contrast agent (iodixanol)

INTERVENTIONS:
Drug: contrast agent (iopromide) — coronary angiography using the allocated contrast agent
  Arms: iopromide
Drug: contrast agent (iodixanol) — coronary angiography using the allocated contrast agent
  Arms: iodixanol

SUMMARY:
In the treatment of coronary heart disease which is the major cause of heart attack, direct mechanical treatment with catheters such as the coronary angiography, coronary balloon intervention and stenting intervention are the mainstay of therapy in recent years. In that procedures, the investigators should use the contrast media, and it may cause kidney toxicity especially in the patients with underlying kidney disease and decreased kidney function. The investigators intended to find out which contrast agent has less kidney toxicity in the catheter based treatment of coronary arterial diseases in patients with underlying decreased kidney function

DETAILED DESCRIPTION:
Iodixanol, a nonionic, dimeric, iso-osmolar contrast medium (IOCM), may be less nephrotoxic than nonionic, monomeric, low-osmolar contrast media (LOCMs) in high-risk patients. We compared the nephrotoxicity of iodixanol with that of iopromide, an nonionic, monomeric LOCM, in patients with renal impairment.

ELIGIBILITY:
Inclusion Criteria:

* patients who undergo coronary catheterization
* creatinine clearance rates ≤ 60 mL/min using the Cockcroft-Gault formula

Exclusion Criteria:

* pregnancy or lactation
* having received contrast media within 7 days of study entry
* emergent coronary angiography
* acute renal failure or end-stage renal disease requiring dialysis
* history of hypersensitivity reaction to contrast media
* unstable hemodynamic states such as cardiogenic shock, pulmonary edema or needing mechanical ventilation
* multiple myeloma
* parenteral use of diuretics
* use of N-acetylcysteine
* use of metformin or nonsteroidal anti-inflammatory drugs within 48 hours of the procedure

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 420 (Estimated)
Dates: Start 2009-02; Primary Completion 2010-05 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Incidence of contrast induced nephropathy, defined as either a relative increase in serum creatinine from baseline of >=25% or an absolute increase of >=0.5mg/dL(44.2µmol/L) | days 1 and 2

SECONDARY OUTCOMES:
proportion of patients exhibiting an increase in serum creatinine of >=0.5mg/dL(44.2µmol/L), the proportion with a >=1.0 mg/dL(88.4µmol/L) increase in serum creatinine, and the mean peak increase in serum creatinine | days 1 and 2

CONTACTS AND LOCATIONS:
Overall Officials: Tae-Jin Youn, MD, PhD, Study Director — Facility: Cardiovascular Center, Seoul National University Bundang Hospital
Locations (1):
- Cardiovascular Center, Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea